CLINICAL TRIAL: NCT04234971
Title: Cost Effectiveness in Alveolar Bone Grafting in Patients with Cleft Lip and Palate: a Randomized Clinical Trial
Brief Title: Cost Effectiveness in Alveolar Bone Grafting in Patients with Cleft Lip and Palate
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Matthew Greives, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HSC-MS-19-1027
Record Dates: First submitted 2020-01-15; First posted 2020-01-21 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Cleft Lip and Palate
Keywords: alveolar bone graft; Bone Morphogenic Protein; Demineralized Bone Matrix; cleft lip
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To prevent surgeon bias in operative time and therefore cost, randomization assignments will be concealed at the beginning of surgery. The surgeon will start with closure of the oronasal fistula first. Once that is completed, the envelope will be opened and reveal the type of bone graft selected. The surgeon will then either harvest the additional ICBG or open the packets for the DBM/BMP and pack the selected type of bone into the alveolus.
  Outcomes assessor including orthodontist and clinical research evaluator will be blinded to treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (DBM/BMP) (Experimental): Patient undergoes Alveolar bone graft with DBM/BMP
  Interventions: Drug: Intervention group (DBM/BMP)
- Control group(autologous ICBG) (Active Comparator): Patient undergoes Alveolar Bone Graft with Iliac Crest Bone graft.
  Interventions: Drug: Control group(autologous ICBG)

INTERVENTIONS:
Drug: Intervention group (DBM/BMP) — All patients will undergo a standard procedure for exposure of the cleft alveolar defect and closure of all oronasal fistulae. After induction of general anesthesia, the patient will be intubated with an oral ray tube and prepped and draped in sterile fashion. Pre-operative antibiotics will be given to cover oral flora (i.e. Unasyn or clindamycin if penicillin allergy exists). The intra-oral space will be exposed and the nasal floor and palatal mucosa will be primarily closed to create a water-tight space for the graft. The integrity of the nasal floor mucosa will be tested using methylene blue dye. Following closure of the fistula, the alveolar bone graft will be performed. For the treatment group, 10cc of crushed DBM will be mixed with the micro-sized sponge of rh-BMP-2 (Infuse Bone Graft, Medronic, Minneapolis, MN). The sponge and DBM will then be packed into the defect to completely fill the bony space (FIGURE 3). The anterior mucosa will then be closed.
  Arms: Intervention group (DBM/BMP)
Drug: Control group(autologous ICBG) — The patient will be induced with anesthesia, prepped, and draped. The intra-oral space will be exposed and the nasal floor and palatal mucosa will be primarily closed to create a water-tight space for the graft. The integrity of the nasal floor mucosa will be tested using methylene blue dye. Following closure of the fistula, the alveolar bone graft will be performed.In the control group, the ICBG will be harvested percutaneously using the Accumed bone graft harvesting system. Briefly, an incision will be made in iliac crest and drill bit inserted. Multiple passes of the drill be used to harvest as much autograft bone as possible from the cancellous region of the iliac crest.Following harvest, fibrin glue will be instilled for hemostasis and a Ropivicaine On-Q pain pump inserted for post-operative pain control. The harvest bone graft will be packed into the alveolar defect in a similar fashion and the mucosa closed anteriorly.
  Arms: Control group(autologous ICBG)

SUMMARY:
The purpose of this trial is to evaluate if the use of Bone Morphogenic Protein(BMP)/Demineralized Bone Matrix (DBM) versus the use of autologous Iliac Crest Bone Graft (ICBG) will result in an increase in total cost effectiveness for patients undergoing alveolar bone graft (ABG) for Cleft Lip and Palate (CLP) and to see if patients who are treated with DBM/BMP will have reduced post-operative pain scores,reduced operative times,and similar rates of bone healing compared to conventional ICBG.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CLP(unilateral or bilateral)
* Radiographically evident open bone defect of the alveolus
* Dentition evaluated by orthodontist and cleared for ABG surgery

Exclusion Criteria:

* Patients without CLP
* Previous failed repair of alveolar cleft
* Patients who have previously undergone successful ABG
* Patients without an alveolar defect
* Patients whose parents refuse to consent to randomization
* Patients who have a syndromic CLP

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Health system costs per successful bone graft. | One year post graft
  Health system costs will be reported as the total sum of all costs including incremental surgeon time costs, hospital costs, revision costs, and additional outpatient costs for clinic or ER visits. Bone graft success be defined as no need for a repeat bone graft, as well as by assessment by blinded orthodontist evaluations of the Post op Cone beam computed tomography(CBCT).

SECONDARY OUTCOMES:
Graft Success | 3 months post graft
  Graft success as indicated by number of patients that did not have exposure of graft as assessed by post op CBCT
Infection | 3 months post graft
  Graft success as indicated by number of patients that had no graft infection as assessed by post op CBCT
Fistula Recurrence | 3 months post graft
  Graft success as indicated by number of patients that had no recurrence of oronasal fistula as assessed by post op CBCT
Rate of Revision ABG | 3 months post graft
  Graft success as indicated by number of patients that had no no need for repeat bone graft as assessed by post op CBCT
Operative Time | 1 day
  Total time for operation
Anesthesia Time | 1 day
  total time of anesthesia
Post Operative Pain Scores | 1 week post operatively
  Change in pain as assessed by the numeric Rating Scale(NRS) for pain. The NRS total score ranges form 0(no hurt) to 10(hurts worst)
Pain Medication Usage | 1 week post operatively
  Total dose of post-operative narcotics used
Post Op Fever | 3 months
  Number of patients with the post operative complication fever
Drainage from Fistula | 3 months
  Number of patients with the post operative complication drainage from donor site or alveolar site
Post Op ER Visits | 3 months.
  Number of patients with the post operative complication ER or primary care visits

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Greives, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No